CLINICAL TRIAL: NCT05176509
Title: A Multicenter, Open-Label, Phase I Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of the Combination of YH003, YH001 and Pembrolizumab in Subjects with Advanced Solid Tumors
Brief Title: A Study to Evaluate the Combination of YH003, YH001 and Pembrolizumab in Subjects with Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eucure (Beijing) Biopharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YH003005
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Solid Tumor
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention/treatment (Experimental)
  Interventions: Drug: YH003; Drug: YH001; Drug: Pembrolizumab

INTERVENTIONS:
Drug: YH003 — YH003 will be administered intravenously over 60 minutes every 21-day cycle.
Drug: YH001 — YH001 will be administered intravenously over 60 minutes every 21-day cycle.
Drug: Pembrolizumab — Pembrolizumab will be administered intravenously over 30 minutes every 21-day cycle.

SUMMARY:
A Multicenter, Open-Label, Phase I Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of the Combination of YH003, YH001 and Pembrolizumab in Subjects with Advanced Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects must have the ability to understand and willingness to sign a written informed consent document.
* 2. Subjects must have histologically advanced or cytologically confirmed solid tumor.
* 3. Subjects have progressed on after treatment with at least one standard therapy, or intolerant of the standard therapy, or no standard therapy accessible to the patients due to any reason
* 4. Subject must have at least 1 unidimensional measurable disease by RECIST 1.1(Eisenhauer et al., 2009).
* 5. Subjects must be age 18 years or older.
* 6. Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* 7. Life expectancy ≥3 months based on investigator's judgement.
* 8. Subjects must meet the following laboratory values at the screening
* 9. Women of reproductive potential must have negative serum beta human chorionic gonadotropin (β -HCG) pregnancy test within 7 days of the first dose of study drugs.
* 10. Women of reproductive potential who are sexually active with a non-sterilized male must consistently use highly effective contraception/birth control between signing of the informed consent and 120 days after the last administration of the study drugs.

Exclusion Criteria:

* 1. Subjects have another active invasive malignancy within 5 years
* 2. Subjects must not have received any anticancer therapy or another investigational agent within the longer of 4 weeks or 5 half-lives before the first dose of the study treatment
* 3. Subjects with a history of ≥ Grade 3 immune-related adverse events resulted from previous immunotherapy.
* 4. History of clinically significant sensitivity or allergy to monoclonal antibodies and their excipients or known allergies to antibodies produced from Chinese hamster ovary cells, which in the opinion of the Investigator suggests an increased potential for an adverse hypersensitivity to YH003, YH001 or Pembrolizumab.
* 5. Primary central nervous system (CNS) malignancies or symptomatic CNS metastases.
* 6. History of (non-infectious) pneumonitis that required corticosteroids or current pneumonitis, or history of interstitial lung disease.
* 7. Subjects must not have a known or suspected history of an autoimmune disorder
* 8. Clinically uncontrolled intercurrent illness, including active coagulopathy, uncontrolled diabetes, psychiatric illness that would limit compliance with the study requirements and other serious medical illnesses requiring systemic therapies.
* 9. Has an active infection requiring systemic therapy.
* 10. Severe cardiovascular disease including symptomatic congestive heart failure (New York Heart Association class III or IV), unstable angina, uncontrolled hypertension, active coagulopathy, uncontrolled diabetes (blood glucose > 250 mg/dl), uncontrolled peritoneal effusion, cardiac arrhythmia, a history of myocardial infarction within 6 months or a history of arterial thromboembolic event and pulmonary embolism within 3 months of the first dose of investigational agent.
* 11. QTcF> 480 ms at baseline; no concomitant medications that would prolong the QT interval; no family history of long QT syndrome.
* 12. Subjects must not have active infection of human immunodeficiency virus (HIV), hepatitis B, hepatitis C or Covid-19.
* 13. Subjects must not have a history of primary immunodeficiency.
* 14. Subjects from endemic area will be specifically screened for tuberculosis. Subjects with active tuberculosis are excluded. Subjects who have received BCG vaccination may have a false positive PPD test. These subjects are eligible if they have a negative Interferon Gamma Release Assay (IGRA).
* 15. Subjects must not receive concurrent or prior use of an immunosuppressive agent within 4 weeks of the first dose
* 16. Major surgery within 4 weeks prior to study entry and Minor surgery within 2 weeks prior to the first dose.
* 17. Subjects must not have received any vaccine within 28 days before the first dose, and subjects, if enrolled, should not receive live vaccines during the study or for 180 days after the last dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | up to 1 year after the last dosing
  The safety will be assessed by monitoring the adverse events (AE) per NCI CTCAE v5.0
Maximum tolerated dose (MTD) and/or Recommended phase 2 dose (RP2D) | up to 1 year after the last dosing
  The MTD and/or RP2D will be determined based on the data of safety and tolerability

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Blacktown Cancer and Haematology Centre, Clinical Trials, Block C, Level 3, 18 Blacktown Road, Blacktown, New South Wales
  - "Oncology Clinical Trial Unit St George Private Hospital 1 South Street", Kogarah, New South Wales
  - 55 Commercial Rd, Level 2 WBRC, Melbourne, Victoria
  - Level 3, Suite 7, North Building, Frankston Private, 5 Susono Way, Frankston, Prahran, Victoria